CLINICAL TRIAL: NCT03805932
Title: A Phase I Study of Moxetumomab Pasudotox-tdfk (Lumoxiti (TM)) and Either Rituximab (Rituxan (R)) or Ruxience for Relapsed Hairy Cell Leukemia
Brief Title: Moxetumomab Pasudotox-tdfk (Lumoxiti(TM)) and Either Rituximab (Rituxan(R)) or Ruxience for Relapsed Hairy Cell Leukemia
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Robert Kreitman, M.D., Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 190042; 19-C-0042
Record Dates: First submitted 2019-01-15; First posted 2019-01-16 (Actual); Results first posted 2023-11-28 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Hairy Cell Leukemia
Keywords: HCL Variant; Recombinant Immunotoxin; Monoclonal Antibody; Targeted Therapy; Biologic Therapy
MeSH Terms: conditions — Leukemia, Hairy Cell | interventions — immunotoxin HA22; Rituximab; Dexamethasone; Calcium Dobesilate; Acetaminophen; Diphenhydramine; Famotidine; Aspirin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Moxetumomab - Dose Escalation 30 mcg/kg (Experimental): Arm 1 Moxetumomab Pasudotox-tdfk + Rituximab
  Interventions: Drug: Moxetumomab Pasudotox-tdfk; Biological: Rituximab; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Famotidine; Drug: Aspirin
- Moxetumomab - Dose Expansion 40 mcg/kg (Experimental): Arm 1 and Arm 2 Moxetumomab Pasudotox-tdfk + Ruxience
  Interventions: Drug: Moxetumomab Pasudotox-tdfk; Biological: Ruxience; Drug: Dexamethasone; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Famotidine; Drug: Aspirin

INTERVENTIONS:
Drug: Moxetumomab Pasudotox-tdfk — Moxetumomab pasudotox-tdfk is administered at 30-40 ug/Kg intravenous (iv) over 30 min given on days 1, 3, 5 of each cycle.
  Other Names: Lumoxiti
Biological: Rituximab — Rituximab will be administered at 375mg/m^2 intravenous (iv), 50-400 mg/hour (hr). On cycle 1, Rituximab is given on day -2, on subsequent cycles, Rituximab is given on day 1.
  Other Names: Rituxan
  Arms: Moxetumomab - Dose Escalation 30 mcg/kg
Biological: Ruxience — Ruxience will be administered at 375mg/m^2 intravenous (iv), 50-400 mg/hour (hr). On cycle 1, Ruxience is given on day -2, on subsequent cycles, Ruxience is given on day 1 (Delta)
  Other Names: Rituximab-pvvr
  Arms: Moxetumomab - Dose Expansion 40 mcg/kg
Drug: Dexamethasone — 12 mg Cycle 1, Day -2; Cycles 2-8, Day 1. Administer 0.5-2 hours before rituximab/Ruxience. If participant has previous reaction to rituximab/Ruxience, give 12mg. If participants tolerate rituximab/Ruxience without problems, may hold at discretion of provider. Pre-medications are given prior to rituximab/Ruxience on day 1.
  Other Names: Ozurdex; Maxidex; DexPak 6 Day
Drug: Acetaminophen — 650 mg Cycle 1, Day -2, Day 1, Day 3, Day 5. To be given 30-90 minutes prior to every moxetumomab pasudotox-tdfk infusion and recommended every 6 hours x 4 after the end of infusion; Cycles 2-8, Day 1, Day 3, Day 5. To be given 30-90 minutes prior to every moxetumomab pasudotox-tdfk infusion and recommended every 6 hours x 4 after the end of infusion. Pre-medications are given prior to rituximab/Ruxience on day 1.
  Other Names: Tylenol; Ofirmev; FeverAll
Drug: Diphenhydramine — 25-50 mg Cycle 1, Day -2; Cycles 2-8, Day 1. Pre-medications are given prior to rituximab/Ruxience on day 1. May be given prior to moxetumomab pasudotox-tdfk at discretion of principal investigator.
  Other Names: Benadryl; Nytol; Banophen
Drug: Famotidine — 20-40 mg Cycle 1, Day -2; Day 1, Day 3, Day 5. To be given 30-90 minutes prior to every moxetumomab pasudotox-tdfk infusion and is recommended every 12 hours x 2 after the end of infusion; Cycles 2-8, Day 1, Day 3, Day 5. To be given 30-90 minutes prior to every moxetumomab pasudotox-tdfk infusion and is recommended every 12 hours x 2 after the end of infusion. Pre-medications are given prior to rituximab/Ruxience on day 1.
  Other Names: Pepcid AC; Pepcid; Acid Controller
Drug: Aspirin — 81 mg Cycle 1, Days 1-8; Cycles 2-8, Days 1-8. Only if platelet counts ≥ 100 x 109/L.
  Other Names: Ecotrin; Enteric Coated Aspirin; Buffered Aspirin

SUMMARY:
Background:

Hairy cell leukemia (HCL) is a rare, slow-growing blood cancer in which the bone marrow makes too many of certain white blood cells. The antibody Rituximab/Ruxience binds to a protein in cancerous white blood cells and is often used to treat HCL. Researchers want to see if combining it with the drug Moxetumomab pasudotox-tdfk (also called Lumoxiti) can fight HCL better.

Objective:

To test the safety of Moxetumomab pasudotox taken with Rituximab/Ruxience for people with HCL or HCL variant.

Eligibility:

People age 18 years and older with HCL or HCL variant that has not responded to standard therapy

Design:

Participants will be screened with:

Medical history

Physical exam

Blood, heart, and urine tests

Test of blood oxygen levels

Review of bone marrow. This can be from previous test results or a new sample.

Scans

Exercise test

Participants will get the study drugs in up to 8 cycles. A cycle will last about 28 days.

The study drugs will be given through a plastic tube in a vein.

In the first week of cycle 1, participants will have:

1 visit to get Rituximab or Ruxience for 7.5 hours

3 visits to get Lumoxiti for 30 minutes per infusion

In the first week of cycles 2-8, participants will have:

1. visit to get Rituximab/Ruxience for 2-4 hours and Lumoxiti for 30 minutes
2. visits to get Lumoxiti for 30 minutes per infusion

Participants will be asked to drink lots of water and take aspirin during the cycles. They will get drugs to minimize allergic reactions.

Participants will repeat screening tests at visits throughout the cycles and 1 follow-up visit. They may have an eye exam.

...

DETAILED DESCRIPTION:
Background:

* Hairy cell leukemia (HCL) is an indolent cluster of differentiation-22 (CD22+) B-cell leukemia comprising 2% of all leukemias, or approximately 1200 of the 62,130 new cases of leukemia/year in the United States (US). HCL variant (HCLv), also CD22+, is 10-20% as common as HCL, but more common in the relapsed/refractory population due to its poor prognosis and response to standard purine analog chemotherapy. hairy cell leukemia variant (HCL-V) cells are cluster of Differentiation 25 (CD25)-negative and wild type for BRAF, so HCLv patients are not candidates for BRAF inhibitors. CD25+ classic-appearing HCL-cells that express unmutated IGHV4-34 (Immunoglobulin Heavy Variable 4-34) are wild-type for BRAF, remain brightly CD22 positive, and confer a poor prognosis when treated with chemotherapy.
* Moxetumomab pasudotox-tdfk is a recombinant immunotoxin containing a variable domain (Fv) fragment of an anti-CD22 monoclonal antibody and truncated Pseudomonas exotoxin, which kills CD22+ cells by binding to CD22 via the (Fv) fragment, and induction of apoptotic cell death catalytic inhibition of protein synthesis in the cytosol.
* Moxetumomab pasudotox-tdfk in phase 1 testing demonstrated a high complete response (CR) rate in patients with chemoresistant HCL, without dose-limiting toxicity (DLT), but with reversible grade 2 hemolytic uremic syndrome (HUS) not requiring plasmapheresis.
* Moxetumomab pasudotox-tdfk completed multicenter phase 3 testing in 80 patients, meeting its complete response (CR) endpoint, with 8.8% incidence each of capillary leak syndrome (CLS, grade 3-4 2.5%), and HUS (grade 3-4 6.3%), both reversible.
* Moxetumomab pasudotox-tdfk is the only known non-chemotherapy-containing regimen for HCL which can consistently eradicate minimal residual disease (MRD), and this is associated with prolonged CR durations. Recently, US Food and Drug Administration (FDA) has accepted the Biologics License Application (BLA) for moxetumomab pasudotox-tdfk as the treatment of adult patients with HCL.
* Patients who did not achieve CR, or CR with MRD, often made neutralizing antibodies to the bacterial-based toxin, and/or had collections of HCL cells not completely eradicated by Moxetumomab pasudotox-tdfk. Both issues may be addressed by the addition of anti-cluster of differentiation 20 (CD20) monoclonal antibody (Mab) rituximab or Ruxience to Moxetumomab pasudotox-tdfk.

Objective:

-To determine the safety and toxicity of Moxetumomab pasudotox-tdfk and rituximab/Ruxience used at the planned dose level, in patients with HCL and HCLv.

Eligibility:

* HCL or HCLv with at least 1 prior purine analog, and, for HCL patients with >=2-years 1 month response, at least 1 other therapy.
* Need for treatment, either 1) absolute neutrophil count (ANC) <1/nL, 2) hemoglobin (Hgb) <10g/dL, 3) platelet (Plt) <100/nL, 4) symptomatic splenomegaly, or enlarging HCL mass > 2cm in short axis
* Serum creatinine < 1.5 mg/dL, or creatinine clearance greater than or equal to 60 mL/min by Cockcroft-Gault equation, where creatinine clearance = (140-age)(kg weight)/(72 x Creatinine).
* No uncontrolled infection or cardiopulmonary dysfunction

Design:

* Phase I trial, two arm, non-randomized, dose escalation
* Administration:

  * Patients 1-13: Moxetumomab pasudotox-tdfk 30-40 mcg/kg intravenous (iv) over 30 min, Rituximab 375 mg/m^2 iv, 50-400 mg/hr.
  * Patients 14-26: Moxetumomab pasudotox-tdfk 40 mcg/kg intravenous (iv) over 30 min, Ruxience 375 mg/m2 iv, 50-400 mg/hr
  * Rituximab or Ruxience day 1 (begin day -2 on cycle 1), Moxetumomab pasudotox-tdfk days 1, 3, and 5.
  * Patients will receive up to 4 cycles past documentation of CR without MRD, maximum 8.
  * To prevent renal toxicity and hypovolemia, patients will be encouraged to drink water gradually, approximately 0.5-1 cup/hour or 6L/day, not going >3 hours without drinking from days 1 to 8 and to keep a hydration diary to record daily fluid consumption.
  * To prevent rituximab/Ruxience toxicity, patients will receive prophylactic dexamethasone orally 0.5- 2 hours before the 1st dose of rituximab, and before subsequent doses until rituximab/Ruxience infusion reactions are not seen. Patients will also receive diphenhydramine, famotidine, and acetaminophen.
  * Dexamethasone 4 mg orally (maximum 2 doses/day) will be given as needed to treat nausea or fever associated with Moxetumomab pasudotox-tdfk, which might prevent adequate water intake
* Statistical design:

  * Up to 26 patients are intended to be treated in the trial. While a total of 26 evaluable patients will be enrolled, the accrual ceiling will be set at 30 to include screen failures and inevaluable patients.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Diagnosis of hairy cell leukemia (HCL) or Hairy cell leukemia variant (HCLv).
* Treatment required for either 1) Absolute neutrophil count (ANC) <1/nL, 2) Hemoglobin <10g/dL, 3) Platelets<100/nL, 4) symptomatic splenomegaly, or 5) enlarging HCL mass > 2cm in short axis. Patients who have eligible blood counts within 4 weeks from the initiation of study will not be considered ineligible if subsequent blood counts prior to enrollment fluctuate and become ineligible up until the time of enrollment.
* Patients must be Pseudomonas-immunotoxin naive.
* HCL or HCLv with at least 1 prior purine analog, and, for HCL patients with >=2-years 1 month response, at least 1 other therapy. Age greater than or equal to 18 years as the disease under study, HCL/HCLv, has not been reported in children < age 18.
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to2 (Karnofsky greater than or equal to 60%)
* Patients must have adequate organ and marrow function as defined below:

  * Total bilirubin less than or equal to 1.5 mg/dL, unless consistent with Gilbert's (ratio between total and direct bilirubin > 5)
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) less than or equal to 3x upper limit of normal (ULN)
  * Alkaline phosphatase < 2.5 ULN
  * Serum creatinine less than or equal to 1.5 mg/dL or creatinine clearance greater than or equal to 60 mL/min by Cockcroft-Gault equation, where creatinine clearance = (140-age)(Kg weight)/(72 x Creatinine)
  * Serum albumin greater than or equal to 2 g/dL
  * Partial thromboplastin time (PTT) or Prothrombin time (PT)/International Normalized Ratio < 2.5x ULN (If on warfarin, PT/INR < 3.5x ULN; If on any other anticoagulation, Prothrombin time (PT) < 2.5x baseline)
  * Fibrinogen greater than or equal to 0.5 lower limit of normal
* The effects of moxetumomab pasudotox-tdfk and rituximab/Ruxience on the developing human fetus are unknown therefore participants must use effective methods of contraception as directed below.

  * Females of childbearing potential (< 50 years) who are sexually active with a non-sterilized male partner must use a highly effective method of contraception prior to study entry and or the duration of study participation and must agree to continue using such precautions for 12 months after completion of rituximab/Ruxience administration. Contraception after this point should be discussed with a responsible physician. Periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of contraception. Females of childbearing potential are defined as those who are not surgically sterile (i.e., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or those who are premenarchal or postmenopausal (defined as 12 months with no menses without an alternative medical cause). A highly effective method of contraception is defined as one that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Not all methods of contraception are highly effective. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately.
  * Non-sterilized males who are sexually active with a female partner of childbearing potential must use an effective method of contraception from Day 1 until 90 days after receipt of the final dose of investigational product. It is required that a female partner of a male subject also use an effective method of contraception throughout this period.
* Ability of subject to understand and the willingness to sign a written informed consent document.
* Patients must be willing to co-enroll in the investigators companion protocol 10C-0066 titled Collection of Human Samples to Study Hairy Cell and other Leukemias, and to Develop Recombinant Immunotoxins for Cancer Treatment.

EXCLUSION CRITIERIA:

* Patients who have had chemotherapy, immunotherapy or radiotherapy within 4 weeks or treatment with rituximab/Ruxience within last 3 months prior to initiation of treatment.
* Patients who are receiving any other investigational agents.
* Breastfeeding within the projected duration of the study, starting with the screening visit through 6 months after the last dose of rituximab/Ruxience. Pregnant women are excluded from this study because moxetumomab pasudotox-tdfk and rituximab/Ruxience are agents with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with moxetumomab pasudotox-tdfk and rituximab/Ruxience, breastfeeding should be discontinued if the mother is treated with moxetumomab pasudotox-tdfk and rituximab/Ruxience.
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, uncontrolled pulmonary infection, pulmonary edema or psychiatric illness/social situations that would limit compliance with study requirements.
* Patients with retinal or choroidal detachment.
* Positive for Hepatitis B core antibody or surface antigen unless the patient is on Tenofovir or Entecavir and Hepatitis B Viral deoxyribonucleic acid (DNA) load is <2000 IU/mL
* Active second malignancy requiring treatment other than minor resection of indolent cancers like basal cell and squamous skin cancers.
* Human immunodeficiency virus (HIV)-positive patients unless taking appropriate anti-HIV medications with a cluster of differentiation 4 (CD4) count of > 200. Otherwise, there may be an increased risk of lethal infections when temporarily suppressing normal B-cells.
* History of an allogeneic bone marrow transplant.
* Patients with a history of both thromboembolism and known congenital hypercoagulable conditions.
* Radioimmunotherapy within 2 years prior to enrollment in the study.
* Patients with history of thrombotic microangiopathy or thrombotic microangiopathy/hemolytic uremic syndrome (HUS).
* Patients with corrected QT interval (Frederica) elevation > 500 msec (manually over-read by medically qualified person) based on at least two separate 12-lead ECGs.
* Patients on high dose estrogen (defined as > 0.625 mg/day of an estrogen compound).
* Oxygen saturation at rest < 88% measured by pulse oximetry or partial pressure of oxygen (PaO2) less than or equal to 55 mm Hg.
* Patients with life expectancy of less than 6 months.
* Patients with clinical evidence of disseminated intravascular coagulation (Grade 3-4).
* Patients with < 50% of predicted forced expiratory volume (FEV1) or < 50% of predicted diffusing capacity for carbon monoxide, corrected for hemoglobin concentration and alveolar volume (DLCO). Note: Patients with no prior history of pulmonary illness are not required to have pulmonary function testing (PFT). Forced expiratory volume will be assessed after bronchodilator therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Kreitman, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All individual participant data (IPD) recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to Biomedical Translational Research Information System (BTRIS) and with the permission of the study principal investigator (PI).

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2019-C-0042.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Moxetumomab - Dose Escalation 30 mcg/kg: Participants with Relapsed/Refractory Hairy Cell Leukemia (HCL) or Hairy Cell Leukemia (HCLv)
  Arm 1 Moxetumomab Pasudotox-tdfk + Rituximab
  Dose escalation treatment with moxetumomab -pasudotox-tdfk and rituximab Moxetumomab pasudotox-tdfk is administered at 30 ug/Kg intravenous (iv) over 30 min given on days 1, 3, 5 of each cycle.
  Rituximab will be administered at 375mg/m^2 iv, 50-400 mg/hour (hr). On cycle 1, Rituximab is given on day -2, on subsequent cycles, Rituximab is given on day 1.
- Moxetumomab - Dose Expansion 40 mcg/kg: Dose expansion; treatment with moxetumomab -pasudotox-tdfk and Ruxience
  Arm 1 and Arm 2 Moxetumomab Pasudotox-tdfk + Ruxience
  Moxetumomab pasudotox-tdfk is administered at 40 ug/Kg intravenous (iv) over 30 min given on days 1, 3, 5 of each cycle.
  Ruxience will be administered at 375mg/m^2 iv, 50-400 mg/hour (hr). On cycle 1, Ruxience is given on day -2, on subsequent cycles, Ruxience is given on day 1 (Delta)
Period: Overall Study
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg
Started | 3 | 15
Completed | 3 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Moxetumomab - Dose Escalation 30 mcg/kg: Participants with Relapsed/Refractory Hairy Cell Leukemia (HCL) or Hairy Cell Leukemia (HCLv)
  Arm 1 Moxetumomab Pasudotox-tdfk + Rituximab
  Dose escalation treatment with moxetumomab -pasudotox-tdfk and rituximab Moxetumomab pasudotox-tdfk is administered at 30-40 ug/Kg intravenous (iv) over 30 min given on days 1, 3, 5 of each cycle.
  Rituximab will be administered at 375mg/m^2 iv, 50-400 mg/hour (hr). On cycle 1, Rituximab is given on day -2, on subsequent cycles, Rituximab is given on day 1.
- Moxetumomab - Dose Expansion 40 mcg/kg: Dose expansion; treatment with moxetumomab -pasudotox-tdfk and Ruxience
  Arm 1 and Arm 2 Moxetumomab Pasudotox-tdfk + Ruxience
  Moxetumomab pasudotox-tdfk is administered at 30-40 ug/Kg intravenous (iv) over 30 min given on days 1, 3, 5 of each cycle.
  Ruxience will be administered at 375mg/m^2 iv, 50-400 mg/hour (hr). On cycle 1, Ruxience is given on day -2, on subsequent cycles, Ruxience is given on day 1 (Delta)
- Total: Total of all reporting groups
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg | Total
Number analyzed (Participants) | 3 | 15 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 10 | 11
  >=65 years | 2 | 5 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.17 (8.98) | 60.07 (8.64) | 60.25 (8.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 14 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 15 | 18
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 14 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 15 | 18

OUTCOME MEASURES:

1. Primary Outcome: Recommended Safe Dose of Moxetumomab Pasudotox-tdfk
Description: Recommended safe dose of moxetumomab pasudotox-tdfk is defined as the treatment of 10 participants with no more than 2 experiencing a dose-limiting toxicity (DLT). A DLT is defined as all treatment related Grade 3-5 adverse events (AEs) occurring from the initiation of moxetumomab pasudotox-tdfk therapy to within 30 days after the last dose of moxetumomab pasudotox-tdfk treatment assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 4 weeks
Measure: Number; unit: mcg/kg
Groups:
- All Participants: All participants in Group 1 and Group 2 who received at least one dose of Moxetumomab 30-40 mcg/kg.
Arm/Group | All Participants
Number analyzed (Participants) | 18
mcg/kg | 40

2. Primary Outcome: Recommended Safe Dose of Rituximab/Ruxience
Description: Recommended safe dose of rituximab/Ruxience is defined as the treatment of 10 participants with no more than 2 experiencing a dose-limiting toxicity (DLT). A DLT is defined as all treatment related Grade 3-5 adverse events (AEs) occurring from the initiation of moxetumomab pasudotox-tdfk therapy to within 30 days after the last dose of moxetumomab pasudotox-tdfk treatment assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: 4 weeks
Measure: Number; unit: mcg/kg
Arm/Group | All Participants
Number analyzed (Participants) | 18
mcg/kg | 40

3. Secondary Outcome: Number of Participants Whose Cancer Shrinks or Disappears After Treatment
Description: Number of participants whose cancer shrinks or disappears after treatment defined as minimal residual disease. MRD is no hairy cell leukemia (HCL) in the blood and bone marrow aspirate flow determined by immunohistochemistry (IHC) and flow cytometry of blood and bone marrow aspirate.
Time Frame: 28-42 days after day 1 of the last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg
Number analyzed (Participants) | 3 | 15
Participants | 2 | 11

4. Secondary Outcome: Number of Participants Who Are Minimal Residual Disease (MRD)-Free
Description: MRD-free is defined as participants with no hairy cell leukemia (HCL) in the blood and bone marrow aspirate flow determined by immunohistochemistry (IHC) and flow cytometry of blood and bone marrow aspirate.
Time Frame: 28-42 days after day 1 of the last treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg
Number analyzed (Participants) | 3 | 15
Participants | 2 | 11

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time of initial response until documented tumor progression. Response was assessed by the and is defined as an increase in symptoms or >25% decline in hematologic parameters related to disease, based on the judgement of the principal investigator. ≥50% increase in sum of products of perpendicular diameters of evaluable (> 2cm) lymphadenopathy or appearance of new evaluable lymph nodes > 2 cm short axis.
Time Frame: 28-42 days after day 1 of the last treatment.
Reporting Status: Not Posted, anticipated posting 2026-06

6. Other Pre Specified Outcome: Number of Participants With a Dose-limiting Toxicity (DLT)
Description: Dose limiting toxicity (DLT) is defined as all treatment related Grade 3-5 adverse events (AEs) occurring from the initiation of moxetumomab pasudotox-tdfk therapy to within 30 days after the last dose of moxetumomab pasudotox-tdfk treatment. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). Grade 3 is severe, Grade 4 is life-threatening, and Grade 5 is death related to adverse event.
Time Frame: From the initiation of moxetumomab pasudotox-tdfk therapy to within 30 days after the last dose
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg
Number analyzed (Participants) | 3 | 15
Participants | 0 | 0

7. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 13 days for the first group, and 4 months and 3 days for the second group.
Measure: Count of Participants; unit: Participants
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg
Number analyzed (Participants) | 3 | 15
Participants | 3 | 15

ADVERSE EVENTS:
Time Frame: Date treatment consent signed to date off study, approximately 11 months and 13 days for the first group, and 4 months and 3 days for the second group.
Arm/Group | Moxetumomab - Dose Escalation 30 mcg/kg | Moxetumomab - Dose Expansion 40 mcg/kg
All-Cause Mortality (participants affected / at risk) | 1/3 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/15
Other Adverse Events (participants affected / at risk) | 3/3 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxetumomab - Dose Escalation 30 mcg/kg (N=3) | Moxetumomab - Dose Expansion 40 mcg/kg (N=15)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 1 (1)
Hemolytic uremic syndrome (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxetumomab - Dose Escalation 30 mcg/kg (N=3) | Moxetumomab - Dose Expansion 40 mcg/kg (N=15)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (4)
Alanine aminotransferase increased (Investigations) | 1 (5) | 10 (24)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (2) | 9 (25)
Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (4)
Aspartate aminotransferase increased (Investigations) | 1 (4) | 13 (40)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Bloating (Gastrointestinal disorders) | 1 (1) | 3 (3)
Blood bilirubin increased (Investigations) | 0 (0) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 7 (19)
Blurred vision (Eye disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 2 (5)
CPK increased (Investigations) | 0 (0) | 2 (7)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 4 (6)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Creatinine increased (Investigations) | 0 (0) | 3 (9)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 2 (3)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (2)
Edema face (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 3 (3) | 9 (17)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 1 (2)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (5) | 5 (8)
Fever (General disorders) | 1 (1) | 7 (11)
GGT increased (Investigations) | 0 (0) | 1 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Glucosuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Haptoglobin decreased (Investigations) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 2 (9) | 10 (33)
Hematuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 2 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 8 (17)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperphosphatemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Hypertension (Vascular disorders) | 0 (0) | 5 (13)
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 (0) | 11 (29)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (4)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 7 (16)
Hypophosphatemia (Metabolism and nutrition disorders) | 0 (0) | 6 (20)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 6 (13)
Infusion site extravasation (General disorders) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 5 (5)
Lipase increased (Investigations) | 1 (1) | 1 (7)
Lymphocyte count decreased (Investigations) | 3 (30) | 15 (167)
Lymphocyte count increased (Investigations) | 0 (0) | 1 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (5) | 6 (7)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 6 (22)
Neck edema (General disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 3 (8) | 4 (10)
Pain (General disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
Palpitations (Cardiac disorders) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 1 (1) | 2 (2)
Platelet count decreased (Investigations) | 3 (6) | 13 (28)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Scrotal pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Serum amylase increased (Investigations) | 1 (1) | 1 (2)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 2 (3)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Superficial thrombophlebitis (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 0 (0) | 4 (4)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4)
White blood cell decreased (Investigations) | 3 (9) | 11 (26)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-04-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT03805932/Prot_SAP_002.pdf
  • Informed Consent Form (2025-05-16): https://cdn.clinicaltrials.gov/large-docs/32/NCT03805932/ICF_003.pdf